CLINICAL TRIAL: NCT05327621
Title: A Single Arm, Open-label, Phase II Study to Assess the Efficacy of Pamiparib in Metastatic Castration-Resistant Prostate Cancer Patients With Homologous Recombination Deficiency (HRD) or BRCA1/2 Mutation
Brief Title: Pamiparib in mCRPC With HRD or BRCA1/2 Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHOU FANGJIAN, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-FXY-385
Record Dates: First submitted 2022-03-27; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Metastatic Castration-resistant Prostate Cancer; PARP inhibitor; Homologous Recombination Deficiency; BRCA1/2 Mutation
MeSH Terms: interventions — pamiparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pamiparib (Experimental): Tablets 20mg per os : 40 mg / bid every day in continuous. Patients will be treated with Pamiparib. Cycles are defined in 28-day periods. Disease response will be assessed every 8 weeks (RECIST 1.1). Safety will be assessed continuously.
  Interventions: Drug: Pamiparib

INTERVENTIONS:
Drug: Pamiparib — 40 mg bid per os , 28 day cycle, number of cycles: until progression or unacceptable toxicity develops.
  Other Names: BGB-290

SUMMARY:
The purpose of this study is to assess the efficacy of a PARP inhibitor, Pamiparib, in metastatic castration-resistant prostate cancer patients with homologous recombination deficiency or BRCA 1 or 2 somatic/germline mutation.

DETAILED DESCRIPTION:
This is a single arm, open-label, single center, phase II trial, assessing the efficacy of a PARP inhibitor, Pamiparib, in 50 progressing metastatic castration-resistant prostate cancer patients with at least one line of androgen deprivation therapy or chemotherapy at the metastatic setting, and homologous recombination deficiency or BRCA 1 or 2 somatic or germline mutation.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old, male
2. Have a histologically or cytologically confirmed adenocarcinoma or poorly differentiated carcinoma without neuroendocrine differentiation of the prostate. Mixed histology is accepted, except for small cell carcinoma.
3. Have a deleterious mutation in BRCA1/2 , or HRD score ≥ 9.
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤1
5. BPI<4
6. Metastatic Castration-resistant Prostate Cancer (mCRPC): Presence of measurable target lesion according to RECIST criteria v1.1
7. Male subject has been surgically or medically sterilized and has serum testosterone level ≤1.73nmol/L.
8. Unsterilized male subject uses an acceptable method of contraception (defined as a barrier method with spermicide) to prevent pregnancy during the duration of the study and for 6 months after the last dose of Pamiparib.
9. Experienced disease progression after having received at least 1 prior next-generation androgen receptor-targeted therapies, for metastatic castration-resistant disease.
10. Capable of swallowing the whole capsule.
11. Subjects must have normal organ and bone marrow function at baseline, as defined below:

    Hemoglobin ≥ 9.0 g/dL at least 28 days after transfusion . Absolute neutrophil count ≥ 1.5 × 10^9/L. Platelet count ≥ 100 × 10^9/L. Total bilirubin ≤ 1.5 × the upper limit of normal (ULN) specified. Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase/alanine aminotransferase (ALT) serum glutamic pyruvic transaminase) ≤ 3 × the specified ULN, unless liver metastases are present, in which case it must be ≤ 5 × ULN.
12. Agree to sign informed consent form
13. Agree not to participate in other interventional trials during this trial.

Exclusion Criteria:

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Acute toxicity (CTCAE > grade 2) due to prior cancer therapy.
2. Received chemotherapy, endocrine therapy, biotherapy, radionuclide therapy, immunotherapy, experimental drugs, proprietary anticancer drugs or Chinese herbal medicines within 5 (if known) half-lives or 14 days(if unknown) prior to the first day of taking Pamiparib; For bisphosphonates or approved bone targeting therapy, Pamiparib must be administered at a steady dose for ≥28 days prior to the first day of taking Pamiparib.
3. Received radiation therapy within 21 days.
4. Prior treatment with any PARP inhibitor. Prior chemotherapy with mitoxantrone or platinum-based chemotherapy or cyclophosphamide. Prior treatment with sipuleucel-T or immune check point inhibitors are allowed.
5. Subjects with major surgery within 2 weeks before starting study treatment. Subjects expected to receive major surgery during the trial.
6. Active second malignancy, with the exception of curatively treated non-melanoma skin cancer, carcinoma in situ, or superficial bladder cancer
7. Symptomatic and/or untreated central nervous system metastases
8. Immunocompromised subjects, such as those with positive human immunodeficiency virus (HIV) serology.
9. Subjects with known active hepatitis (e.g. hepatitis B or C).
10. The subject has a serious cardiovascular disease. ( For example, but not limited to: uncontrolled arrhythmia, myocardial infarction)
11. Concomitant use of strong CYP3A inducers or moderate CYP3A inducers . If half-lives is known, a 5 half-lives washout period is required before the start of Pamiparib therapy and a 2-week washout period is required when the half-lives is unknown.
12. History of intolerance to Pamiparib capsule excipients
13. Excluded by investigators

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Radiologic Progression-free Survival (rPFS) | 3 years
  Radiologic progression-free survival will be assessed from the time of the first dose to radiologic disease progression or death from any cause, whichever comes first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From enrollment to primary completion of study (up to approximately 3 years)
  Proportion of patients in complete remission (CR) plus partial remission (PR)
Duration of Response (DOR) | From enrollment to primary completion of study (up to approximately 3 years)
  Time from the start of the first assessment of the tumor as CR or PR to the first assessment of PD (Progressive Disease) or death from any cause.
Time to Response (TTR) | From enrollment to primary completion of study (up to approximately 3 years)
  Time from initiation of treatment to first assessment of tumor as CR or PR.
Clinical Benefit Rate | 3 years
  according to RECIST, is either complete response (CR), partial response (PR) or stable disease (SD) lasting for at least 16 weeks
Prostate Specific Antigen (PSA) Response Rate | From enrollment to primary completion of study (up to approximately 3 years)
  Proportion of patients with a 50% decrease in PSA from baseline
Time to PSA Progression | From enrollment to primary completion of study (up to approximately 3 years)
  Time from initiation of treatment to two consecutive 50% PSA increases from baseline level
Overall Survival (OS) | From enrollment to primary completion of study (up to approximately 3 years)
  Time between the start of treatment and death from any cause
Adverse events | 3 years
  Adverse events are graded according to the CTCAE V4.03

OTHER OUTCOMES:
rPFS stratified by baseline HRD score (HRD score threshold is defined as 9) | 3 years
  The rPFS is defined as the duration from Pamiparib initiation to radiologic disease progression or death from any cause, whichever comes first.
OS stratified by baseline HRD score (HRD score threshold is defined as 9) | 3 years
  The OS is defined as the duration from Pamiparib initiation to any death.

CONTACTS AND LOCATIONS:
Overall Officials: Fangjian Zhou, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China